CLINICAL TRIAL: NCT04095624
Title: Does Preoperative Pain Medication Management Influence Surgical Outcomes in Spinal Fusion: A Randomized Controlled Study
Brief Title: Does Preoperative Pain Medication Management Influence Surgical Outcomes in Spinal Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Serena Hu, Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 47240
Record Dates: First submitted 2019-06-03; First posted 2019-09-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2022-07

CONDITIONS: Opioid Use; Spine Fusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Taper Group (Experimental): Patients randomized to the taper group will have baseline pain score, opioid medication use, and patient reported outcomes 4-6 weeks prior to elective thoracolumbar, lumbar, or lumbosacral spinal fusion surgery. They will receive a scheduled tapering protocol, with a goal of 10-15% reduction in their weekly opioid use, along with weekly phone calls from a study coordinator assessing their ability to taper and pain scores. After surgery, they will receive 6 weekly phone calls from the coordinator, to assess their postoperative opioid medication use and pain scores. At the 6th week phone call, and 3 month and 6 month clinic postoperative clinic visits, they will also repeat patient reported outcome measures.
  Interventions: Behavioral: Spinal Fusion Preoperative Opioid Taper
- Control Group (Active Comparator): Patients randomized to the control group will have baseline pain score, opioid medication use, and patient reported outcomes 4-6 weeks prior to elective thoracolumbar, lumbar, or lumbosacral spinal fusion surgery. They will receive no recommendation or guidance in their preoperative opioid pain medication use, but will received weekly phone calls from a study coordinator assessing their preoperative pain scores. After surgery, they will receive 6 weekly phone calls from the coordinator, to assess their postoperative opioid medication use and pain scores. At the 6th week phone call, and 3 month and 6 month clinic postoperative clinic visits, they will also repeat patient reported outcome measures.
  Interventions: Other: Non-taper Control

INTERVENTIONS:
Behavioral: Spinal Fusion Preoperative Opioid Taper — Guided weekly opioid pain medication reduction via telephone calls prior to elective spinal fusion surgery.
  Arms: Opioid Taper Group
Other: Non-taper Control — Weekly phone calls prior to elective spinal fusion surgery, without opioid pain medication reduction recommendation or guidance.
  Arms: Control Group

SUMMARY:
In light of the current opioid epidemic, there is an urgent need to address chronic opioid use prior to surgery before it is exacerbated by postoperative surgical pain. Our central hypothesis is that patients who taper their opioid use prior to surgery will have reduced postoperative opioid and pain medication usage, less postoperative pain, and improved patient reported outcomes relative to patients that do not taper prior to surgery. Our specific aims include: 1. Determine whether reducing patients' preoperative opioid usage through a structured tapering regimen reduces postoperative opioid and pain medication use. 2. Examine whether reducing patients' preoperative opioid usage through a structured tapering regimen reduces postoperative pain. 3. Determine whether reducing patients' preoperative opioid usage through a structured tapering regimen improves patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Indicated for lumbar, lumbosacral, or thoracolumbar spinal fusion surgery in the departments of Orthopedic Surgery and Neurosurgery
* Daily opioid use for at least 4 weeks prior to the preoperative planning appointment

Exclusion Criteria:

* Suboxone (buprenorphine) use
* Unable to complete patient reported outcome measures (PROMs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Postoperative Opioid Pain Medication Dose | Weekly, month 3, month 6
  Weekly average opioid medication use in morphine equivalent dosage (MED)
Change in Numeric Pain Scale Score | Weekly, month 3, month 6
  Generic measure of average back pain, scale 0-10 with 0 being no pain and 10 being the most pain experienced.
Change from baseline Patient Reported Outcome Measures (PROMs) | Weekly, month 3, month 6
  PROMIS computer adaptive testing: global health, physical function, pain interference, pain behavior, depression, anxiety, fatigue, sleep disturbance, and satisfaction with social roles and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Hu, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baron MJ, McDonald PW. Significant pain reduction in chronic pain patients after detoxification from high-dose opioids. J Opioid Manag. 2006 Sep-Oct;2(5):277-82. doi: 10.5055/jom.2006.0041. PMID 17319259
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Berna C, Kulich RJ, Rathmell JP. Tapering Long-term Opioid Therapy in Chronic Noncancer Pain: Evidence and Recommendations for Everyday Practice. Mayo Clin Proc. 2015 Jun;90(6):828-42. doi: 10.1016/j.mayocp.2015.04.003. PMID 26046416
- [Background] Chu LF, Angst MS, Clark D. Opioid-induced hyperalgesia in humans: molecular mechanisms and clinical considerations. Clin J Pain. 2008 Jul-Aug;24(6):479-96. doi: 10.1097/AJP.0b013e31816b2f43. PMID 18574358
- [Background] Chu LF, Clark DJ, Angst MS. Opioid tolerance and hyperalgesia in chronic pain patients after one month of oral morphine therapy: a preliminary prospective study. J Pain. 2006 Jan;7(1):43-8. doi: 10.1016/j.jpain.2005.08.001. PMID 16414554
- [Background] Crisostomo RA, Schmidt JE, Hooten WM, Kerkvliet JL, Townsend CO, Bruce BK. Withdrawal of analgesic medication for chronic low-back pain patients: improvement in outcomes of multidisciplinary rehabilitation regardless of surgical history. Am J Phys Med Rehabil. 2008 Jul;87(7):527-36. doi: 10.1097/PHM.0b013e31817c124f. PMID 18574345
- [Background] Farrell M. Opiate withdrawal. Addiction. 1994 Nov;89(11):1471-5. doi: 10.1111/j.1360-0443.1994.tb03745.x. PMID 7841858
- [Background] Fishbain DA, Rosomoff HL, Cutler R. Opiate detoxification protocols. A clinical manual. Ann Clin Psychiatry. 1993 Mar;5(1):53-65. doi: 10.3109/10401239309148924. PMID 8394176
- [Background] Heiwe S, Lonnquist I, Kallmen H. Potential risk factors associated with risk for drop-out and relapse during and following withdrawal of opioid prescription medication. Eur J Pain. 2011 Oct;15(9):966-70. doi: 10.1016/j.ejpain.2011.03.006. Epub 2011 May 4. PMID 21546290
- [Background] Mirza SK, Deyo RA, Heagerty PJ, Konodi MA, Lee LA, Turner JA, Goodkin R. Development of an index to characterize the "invasiveness" of spine surgery: validation by comparison to blood loss and operative time. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2651-61; discussion 2662. doi: 10.1097/BRS.0b013e31818dad07. PMID 18981957
- [Background] Nguyen LC, Sing DC, Bozic KJ. Preoperative Reduction of Opioid Use Before Total Joint Arthroplasty. J Arthroplasty. 2016 Sep;31(9 Suppl):282-7. doi: 10.1016/j.arth.2016.01.068. Epub 2016 Mar 17. PMID 27105557
- [Background] Nilsen HK, Stiles TC, Landro NI, Fors EA, Kaasa S, Borchgrevink PC. Patients with problematic opioid use can be weaned from codeine without pain escalation. Acta Anaesthesiol Scand. 2010 May;54(5):571-9. doi: 10.1111/j.1399-6576.2009.02164.x. Epub 2009 Nov 16. PMID 19919582
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Ralphs JA, de C Williams AC, Richardson PH, Pither CE, Nicholas MK. Opiate reduction in chronic pain patients: a comparison of patient-controlled reduction and staff controlled cocktail methods. Pain. 1994 Mar;56(3):279-288. doi: 10.1016/0304-3959(94)90166-X. PMID 8022621
- [Background] Tennant FS Jr, Rawson RA. Outpatient treatment of prescription opioid dependence: comparison of two methods. Arch Intern Med. 1982 Oct;142(10):1845-7. PMID 6181749
- [Background] Townsend CO, Kerkvliet JL, Bruce BK, Rome JD, Hooten MW, Luedtke CA, Hodgson JE. A longitudinal study of the efficacy of a comprehensive pain rehabilitation program with opioid withdrawal: comparison of treatment outcomes based on opioid use status at admission. Pain. 2008 Nov 15;140(1):177-189. doi: 10.1016/j.pain.2008.08.005. Epub 2008 Sep 19. PMID 18804915